CLINICAL TRIAL: NCT05416593
Title: Exploring the Motivational Impact of Individualized Pleasure-Oriented Exercise Sessions in a Health Club Setting: Protocol for a Randomized Controlled Trial
Brief Title: Exploring the Impact of Individualized Pleasure-Oriented Exercise Sessions in a Health Club Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grupo Lusófona (Other)
Responsible Party: Principal Investigator, Diogo Teixeira, Doctor, Grupo Lusófona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GrupoLusofona_RCT_AFFECT
Record Dates: First submitted 2022-05-02; First posted 2022-06-13 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Affect
Keywords: Affect; Affective response; Exercise; Affective determinants; Circumplex model
MeSH Terms: conditions — Motor Activity | interventions — Coe Comfort

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General exercise prescription (FITT) (Placebo Comparator): Exercise group; control; general exercise prescription
  Interventions: Behavioral: General exercise prescription (FITT)
- Affective regulation (AFFECT) (Experimental): Exercise group; experimental; general exercise prescription plus affective response and preferences regulation
  Interventions: Behavioral: Affective regulation (AFFECT)

INTERVENTIONS:
Behavioral: General exercise prescription (FITT) — The (1) control group (FITT) will receive a preexercise evaluation and 3 individualized training sessions based on the ACSM and FITT principles (ACSM, 2021). These are the procedures commonly used for apparently healthy individuals that start to exercise in health clubs.
  Arms: General exercise prescription (FITT)
Behavioral: Affective regulation (AFFECT) — As for the (2) experimental group (AFFECT), the focus will be given to exercise intensity assessment and manipulation. The same preexercise evaluation, number of individualized sessions, and methodological approach (i.e., FITT) will be made. However, individual preferences and experiences regarding exercise intensity will be assessed in the preexercise evaluation. These will be used to select the exercise sessions' initial intensity. Moreover, intensity self-selection guidance and affective response assessments will be made throughout the session for continuous intensity adjustments (aiming for pleasurable feelings).
  Arms: Affective regulation (AFFECT)

SUMMARY:
A call for an exercise prescription aiming at pleasure promotion has been proposed by several authors. This entails that current exercise prescription guidelines are heavily focused on a dose-response relation derived from an effectiveness (e.g., fitness gains) and safety of the prescription (e.g., reduced risk of injury for the general population) standpoint. Despite its relevance, this bipartite or biomedical approach (e.g., rationale for a given dose of a drug and expected outcome) tends to overlook other relevant variables that are needed for, for example, behavior maintenance, or individual preferences. Although some flexibility of this rationale may account for personal differences, how to adequately adjust the training variables to individual characteristics is still poorly explored or even expressed.

The call for a tripartite exercise prescription reflects the bout of evidence that supports the relevance of pleasurable experiences in exercise and their impact on adherence. Thus, besides an effective and safe program, contemplating how to assess and promote exercise-related pleasurable experiences are paramount. As stated in 2011 on the ACSM position stand, affect-regulation did not behold the necessary evidence to be a primary method of exercise prescription, although affect assessment (e.g., through the feeling scale) was proposed to be relevant for exercise intensity self-regulation. A decennial look at the ACSM exercise guidelines shows that although presenting an advancement in affect-related behavioral strategies and theories, no clear indications on operational instruments for assessment and admeasurement of affect are presented depicts a barrier to an adequate advancement in this matter. This can be seen, for example, in ACSM principles for exercise prescription (Frequency, Intensity, Time, and Type; FITT). Although supporting the use of affect regulation for exercise promotion and maintenance, the FITT is not based on a previous (e.g., preexercise evaluation) or in-session affective assessment, and more importantly, does not address how to adjust exercise prescription/supervision aiming to improve the pleasure/displeasure relation.

DETAILED DESCRIPTION:
Background and rationale From a public health standpoint, gyms and health clubs are one of the most relevant contexts of supervised exercise practice, targeting millions of individuals worldwide. However, exercise adherence has proven to be a challenge in the last 20 years. Several indicators show high attrition rates (i.e., clients' dropout in a given period) in these contexts, particularly in the first 6 months.

Individual physical activity promotion can be challenging as it reflects several aspects of a complex human behavior. Many psychological theories and strategies have been used to address this issue, albeit with differentiated results. These are usually based on cognitivist assumptions and have shown small to moderate effects on exercise adherence. However, in recent years, exercise psychology started to shift attention to other constructs that can help expand the predictive value of current theoretical models. Particularly, affective processes (e.g., emotions, mood) have been highlighted as relevant when trying to understand or predict behavior, and a call for a new era - the affectivism - is emerging. This reflects a new parading resulting from decades of evidence in which affective processes can be seen as outcomes, but also as relevant constructs that can expand the understanding of current behavioral strategies and theories.

For example, the latest edition of the American College of Sports Medicine (ACSM) guidelines presented an expanded chapter addressing behavioral theories for increasing physical activity, which, besides the most commonly used (e.g., self-efficacy, self-determination theory, theory of planned behavior), now explores affect regulation as a product of non-conscious motivational processes (e.g., dual-process theories), and the automatic associations between behavior and previous affective response (i.e., remembered affect).

Affective determinants in exercise and the role of exercise intensity

Affect can be understood as an umbrella term that encompasses (1) the most general valenced experiential responses (e.g., pleasure/displeasure; good/bad), termed basic affect or core affect, and (2) emotion and mood, which reflects appraisal processes of basic affect, and are usually called distinct affective states. Several theories and models have been developed in recent years that reflect this conceptualization and the evidence of affect-related constructs, as is the case, for example, of the Affective-Reflective Theory of physical inactivity and exercise (ART); the Physical Activity Adoption and Maintenance (PAAM) model; the Theory of Effort Minimization in Physical Activity (TEMPA), and the Affect and Health Behavior Framework (AHBF).

In the broader look given by the AHBF, the affective response (i.e., how one feels while performing an activity or immediately after completing the activity; core affect), triggers a set of influences that can, via an automatic or reflective affect processing, influence motivation, goals, behavioral intentions and, ultimately, the exercise behavior. As shown in some research, the affective response during exercise has demonstrated to be a determinant of future behavior, and core affective valence and activation the most relevant aspects in this matter. This seems to be grounded in hedonic assumptions (i.e., pursuing pleasure and avoiding displeasure or pain), in which positive (and regular) shifts in affective valence and/or activation tend to increase the likelihood of future exercise behavior, and a negative shift may have an opposite influence.

Regarding exercise characteristics that may influence the affective response, exercise intensity stand out as the most relevant. Current evidence suggests that people present distinct responses as intensity increases. Generally, aerobic activities intensities below the ventilator threshold depict similar patterns among exercisers, given that an increase in intensity usually corresponds to an increase in the pleasurable response. After the ventilator threshold, inter-individual variability marks how soon or accentuated the pleasure decline will be manifested. For resistance training, some evidence also indicates that increases in intensity (e.g., Repetition Maximum (RM) %) are positively associated with pleasure until the 70-80 RM% interval, a moment from which individual characteristics will reflect, albeit unclear at this point at which rate or magnitude, an inverted association with pleasure. Thus, targeting the intensity-pleasure/displeasure relation individually may be of particular relevance for the exercise domain when aiming to promote adherence.

Exercise prescription - a tripartite approach

A call for an exercise prescription aiming pleasure promotion has been proposed by several authors. This entails that current exercise prescription guidelines are heavily focused on a dose-response relation derived from an effectiveness (e.g., fitness gains) and safety of the prescription (e.g., reduced risk of injury for the general population) standpoint. Despite its relevance, this bipartite or biomedical approach (e.g., rationale for a given dose of a drug and expected outcome) tends to overlook other relevant variables needed for, for example, behavior maintenance or individual preferences. Although some flexibility of this rationale may account for personal differences, how to adequately adjust the training variables to individual characteristics is still poorly explored or even expressed.

The call for a tripartite exercise prescription reflects the bout of evidence that supports the relevance of pleasurable experiences in exercise and their impact on adherence. Thus, besides an effective and safe program, contemplating how to assess and promote exercise-related pleasurable experiences are paramount. As stated in 2011 on the ACSM position stand, affect-regulation did not behold the necessary evidence to be a primary method of exercise prescription, although affect assessment (e.g., through the feeling scale) was proposed to be relevant for exercise intensity self-regulation. A decennial look at the ACSM exercise guidelines shows, and although presenting an advancement in affect-related behavioral strategies and theories, that no clear indications on operational instruments for assessment and admeasurement of affect are presented, which depicts a barrier to an adequate advancement in this matter. This can be seen, for example, in ACSM principles for exercise prescription (Frequency, Intensity, Time, and Type; FITT). Although supporting the use of affect regulation for exercise promotion and maintenance, the FITT is not based on a previous (e.g., preexercise evaluation) or in-session affective assessment, and more importantly, does not address how to adjust exercise prescription/supervision aiming to improve the pleasure/displeasure relation.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 45 years old,
* Apparently healthy and without contraindications to exercise,
* Normal weight (BMI ≥18.5 <29.9 Kg/m2);
* To have previous experience in a gym or health club
* To be at least 6 months without any type of regular strength, cardiovascular, or flexibility workouts (< 5 workouts/month) in a health club or any kind of structured sports activity).

Exclusion Criteria:

Before enrollment

* High in the risk stratification for cardiovascular disease (ACSM, 2021)
* High blood pressure (≥ 130/80mmHg) in the initial preexercise evaluation

During the intervention

* Acquired injury
* The inability to perform 2 exercise sessions (48h to 96h apart) in two consecutive weeks

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-11-24 (Actual); Study Completion 2022-11-24 (Actual)

PRIMARY OUTCOMES:
Post-intervention exercise attendance to the health club | During 8 weeks, at day 7, 14, 21, 28, 35, 42, 49, and 56
  Post-intervention weekly exercise frequency, objectively measured by the accesses via the turnstile in the health clubs

SECONDARY OUTCOMES:
Exercise habit measured with the Self-reported behavioral automaticity index (SRBAI) | 5 minutes before the first session
  Automaticity for exercise practice measured with the Self-reported behavioral automaticity index (SRBAI)
Exercise habit measured with the Self-reported behavioral automaticity index (SRBAI) | 5 minutes after the last session
  Automaticity for exercise practice measured with the Self-reported behavioral automaticity index (SRBAI)
Initial behavioral intention to continue exercising; the intention to exercise questionnaire | 5 minutes before the first session
  Behavioral intention as defined by the theory of planned behavior with the intention to exercise questionnaire
Final behavioral intention to continue exercising; the intention to exercise questionnaire | 5 minutes after the last session
  Behavioral intention as defined by the theory of planned behavior with the intention to exercise questionnaire
Motivation to exercise measured with the enjoyment/interest scale of the Intrinsic Motivation Inventory | 5 minutes before the first session
  Intrinsic motivation measured with the enjoyment/interest scale Intrinsic Motivation Inventory
Motivation to exercise measured with the enjoyment/interest scale of the Intrinsic Motivation Inventory | 5 minutes after the last session
  Intrinsic motivation measured with the enjoyment/interest scale Intrinsic Motivation Inventory
Autonomy in exercise practice measured with the perceived choice scale of the Intrinsic Motivation Inventory | 5 minutes before the first session
  Autonomy in exercise practice measured with the perceived choice scale of the Intrinsic Motivation Inventory
Autonomy in exercise practice measured with the perceived choice scale of the Intrinsic Motivation Inventory | 5 minutes after the last session
  Autonomy in exercise practice measured with the perceived choice scale of the Intrinsic Motivation Inventory
Competence in exercise practice measured with the competence scale of the Intrinsic Motivation Inventory | 5 minutes before the first session
  Competence in exercise practice measured with the competence scale of the Intrinsic Motivation Inventory
Competence in exercise practice measured with the competence scale of the Intrinsic Motivation Inventory | 5 minutes after the last session
  Competence in exercise practice measured with the competence scale of the Intrinsic Motivation Inventory
Subjective vitality in exercise measured with the subjective vitality in exercise scale (SVS) | 5 minutes before the first session
  Subjective vitality in exercise measured with the subjective vitality in exercise scale (SVS) as defined by the self-determination theory
Subjective vitality in exercise measured with the subjective vitality in exercise scale (SVS) | 5 minutes after the last session
  Subjective vitality in exercise measured with the subjective vitality in exercise scale (SVS) as defined by the self-determination theory
Feelings in exercise; assessed with the Feeling Scale; score ranges between -5 and +5; higher values represent a better outcome | At minute 5
  Feelings in exercise; assessed with the Feeling Scale; score ranges between -5 and +5; higher values represent a better outcome
Feelings in exercise; assessed with the Feeling Scale; score ranges between -5 and +5; higher values represent a better outcome | At minute 10 of the session
  Feelings in exercise; assessed with the Feeling Scale; score ranges between -5 and +5; higher values represent a better outcome
Feelings in exercise; assessed with the Feeling Scale; score ranges between -5 and +5; higher values represent a better outcome | At minute 15 of the session
  Feelings in exercise; assessed with the Feeling Scale; score ranges between -5 and +5; higher values represent a better outcome
Feelings in exercise; assessed with the Feeling Scale; score ranges between -5 and +5; higher values represent a better outcome | Immediately after resistance exercise
  Feelings in exercise; assessed with the Feeling Scale; score ranges between -5 and +5; higher values represent a better outcome
Feelings in exercise; assessed with the Feeling Scale; score ranges between -5 and +5; higher values represent a better outcome | Immediately after stretching exercise
  Feelings in exercise; assessed with the Feeling Scale; score ranges between -5 and +5; higher values represent a better outcome
Feelings in exercise; assessed with the Feeling Scale; score ranges between -5 and +5; higher values represent a better outcome | At minute 45 of the session
  Feelings in exercise; assessed with the Feeling Scale; score ranges between -5 and +5; higher values represent a better outcome
Feelings in exercise; assessed with the Feeling Scale; score ranges between -5 and +5; higher values represent a better outcome | At minute 50 of the session
  Feelings in exercise; assessed with the Feeling Scale; score ranges between -5 and +5; higher values represent a better outcome
Feelings in exercise; assessed with the Feeling Scale; score ranges between -5 and +5; higher values represent a better outcome | At minute 55 of the session
  Feelings in exercise; assessed with the Feeling Scale; score ranges between -5 and +5; higher values represent a better outcome
Arousal/Activation in exercise; assessed with the Felt Arousal Scale; score ranges between 1 and 6; higher values represent a better outcome | At minute 5
  Activation in exercise; assessed with the Felt Arousal Scale; score ranges between 1 and 6; higher values represent a better outcome
Arousal/Activation in exercise; assessed with the Felt Arousal Scale; score ranges between 1 and 6; higher values represent a better outcome | At minute 10
  Activation in exercise; assessed with the Felt Arousal Scale; score ranges between 1 and 6; higher values represent a better outcome
Arousal/Activation in exercise; assessed with the Felt Arousal Scale; score ranges between 1 and 6; higher values represent a better outcome | At minute 15
  Activation in exercise; assessed with the Felt Arousal Scale; score ranges between 1 and 6; higher values represent a better outcome
Arousal/Activation in exercise; assessed with the Felt Arousal Scale; score ranges between 1 and 6; higher values represent a better outcome | Immediately after resistance exercise
  Activation in exercise; assessed with the Felt Arousal Scale; score ranges between 1 and 6; higher values represent a better outcome
Arousal/Activation in exercise; assessed with the Felt Arousal Scale; score ranges between 1 and 6; higher values represent a better outcome | Immediately after stretching exercise
  Activation in exercise; assessed with the Felt Arousal Scale; score ranges between 1 and 6; higher values represent a better outcome
Arousal/Activation in exercise; assessed with the Felt Arousal Scale; score ranges between 1 and 6; higher values represent a better outcome | At minute 45
  Activation in exercise; assessed with the Felt Arousal Scale; score ranges between 1 and 6; higher values represent a better outcome
Arousal/Activation in exercise; assessed with the Felt Arousal Scale; score ranges between 1 and 6; higher values represent a better outcome | At minute 50
  Activation in exercise; assessed with the Felt Arousal Scale; score ranges between 1 and 6; higher values represent a better outcome
Arousal/Activation in exercise; assessed with the Felt Arousal Scale; score ranges between 1 and 6; higher values represent a better outcome | At minute 55
  Activation in exercise; assessed with the Felt Arousal Scale; score ranges between 1 and 6; higher values represent a better outcome
Initial affective attitudes related to exercise | 5 minutes before the session
  Individual affective attitudes for exercise measured with the Exercise and Me Questionnaire (AFFEXX)
Final affective attitudes related to exercise | 48 hours after the end of the intervention (all sessions)
  Individual affective attitudes for exercise measured with the Exercise and Me Questionnaire (AFFEXX)
Exercise enjoyment measured with the the Physical Activity Enjoyment Scale (PACES) | Measured at baseline; 5 minutes before the session
  Exercise enjoyment measured with the the Physical Activity Enjoyment Scale (PACES)
Exercise enjoyment measured with the the Physical Activity Enjoyment Scale (PACES) | Measured at the end of the intervention (all sessions); 5 minutes after the last session
  Exercise enjoyment measured with the the Physical Activity Enjoyment Scale (PACES)
Anticipated affective response to exercise | 5 minutes before the session
  Anticipated affective response to a future exercise session measured with the Empirical Valence Scale
Final anticipated affective response to exercise | 48 hours after the intervention
  Anticipated affective response to a future exercise session measured with the Empirical Valence Scale
Remembered affect to the previous exercise session | 5 minutes before the session
  Remembered affect of previous exercise session measured with the Visual Analog Scale
Final remembered affect to the previous exercise session | 48 hours after the intervention
  Remembered affect of previous exercise session measured with the Visual Analog Scale

OTHER OUTCOMES:
Resting blood pressure (mmHg) | 10 minutes before the first exercise session
  Resting blood pressure
Heart rate during exercise (bpm) | During all the exercise session (60 minutes); measured in the three sessions
  Heart rate during exercise
Adaption and fatigue to the workout measured with the Hooper index | 24 hours after the session
  Adaption and fatigue to the workout

CONTACTS AND LOCATIONS:
Overall Officials: Diogo S. Teixeira, PhD, Principal Investigator — Grupo Lusófona
Locations (1):
- People Family Club, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teixeira DS, Bastos V, Andrade AJ, Palmeira AL, Ekkekakis P. Individualized pleasure-oriented exercise sessions, exercise frequency, and affective outcomes: a pragmatic randomized controlled trial. Int J Behav Nutr Phys Act. 2024 Aug 5;21(1):85. doi: 10.1186/s12966-024-01636-0. PMID 39103923
- [Derived] Teixeira DS, Ekkekakis P, Andrade AJ, Bastos V, Palmeira AL. Exploring the impact of individualized pleasure-oriented exercise sessions in a health club setting: Protocol for a randomized controlled trial. Psychol Sport Exerc. 2023 Jul;67:102424. doi: 10.1016/j.psychsport.2023.102424. Epub 2023 Mar 15. PMID 37665877